CLINICAL TRIAL: NCT04103411
Title: Effect of High-Intensity Interval Training Compared to Hydrochlorothiazide on Ambulatory Blood Pressure, Cardiovascular Health, Cognition and Mobility in Pre-Hypertensive Older Adults.
Brief Title: Effect of High-Intensity Interval Training Compared to Hydrochlorothiazide on Ambulatory Blood Pressure
Acronym: DIISCCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anil Nigam (Other)
Responsible Party: Sponsor-Investigator, Anil Nigam, MD, cardiologist, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-2319
Record Dates: First submitted 2019-09-18; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Hypertension,Essential; Exercise Activity
MeSH Terms: conditions — Essential Hypertension | interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (HIIT) (Experimental): For the twelve weeks of intervention, participants will have three training sessions per week. Each session will be done on a cycle ergometer and will last approximately 40 minutes. Participants will be supervised by certified kinesiologists and their training programs will be revised every four weeks.
  Interventions: Other: 24h-Ambulatory Blood Pressure
- HydroChloroThiazide (Active Comparator): For this group, participants have to take a diuretic (12,5 mg of Hydrochlorothiazide) daily prescribed by the doctor of this study, for twelve weeks. Participants should also maintain the same lifestyle habits that they had before the study.
  Interventions: Other: 24h-Ambulatory Blood Pressure

INTERVENTIONS:
Other: 24h-Ambulatory Blood Pressure — Effect of High Intensity Interval Training compared to Hydrochlorothiazide on ambulatory Blood Pressure.
  Other Names: Cognition; Cardiovascular Health; Mobility

SUMMARY:
The number of persons with hypertension is increasing and with it the number of related cardiovascular events and related functional or cognitive declines. While studies have suggested that physical activity, in particular, high-intensity interval training (HIIT), could be as efficient as the commonly used antihypertensive medications, no studies have actually compared their effects in the same population. This protocol will determine if HIIT is at least as efficient as hydrochlorothiazide in order to lower 24h-ambulatory blood pressure (BP) in prehypertensive older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age at consent ≥ 60 years;
2. Systolic Blood pressure measured through BPtru™ between SBP ≥ 120 mmHg and < 140 and or DBP ≥ 80 mmHg
3. Being able to sign the informed consent form

Exclusion Criteria:

1. Considered "highly active" according to the International Physical Activity Questionnaire
2. Practicing more than 20 min per week of High-Intensity Interval Training
3. Use of antihypertensive medication
4. Contraindication for the practice of intense physical activity
5. Functional limitations related to the exercise test and to intensive training
6. Cardiovascular pathology
7. Atrial fibrillation
8. Psychiatric or neurological disorder
9. Renal failure
10. MMSE score < 26
11. Persons benefiting of enhanced protection: persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection and patients in emergency situations.
12. Diabetes

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
24h-Ambulatory Blood Pressure | At baseline and after twelve weeks of intervention
  The 24-hour ambulatory measure of the blood pressure (AMBP)

SECONDARY OUTCOMES:
Cardiovascular evaluation | Before and after twelve weeks of intervention
  Maximum incremental cardiopulmonary exercise test (VO2MAX)
Cognitive functions | Before and after twelve weeks of intervention
  Cognitive functions will be measured at rest with a pen-paper battery test by a neuropsychologist. The investigators will measure change of score to the cognitive tests.
Flow Mediated Dilatation (FMD) | Before and after twelve weeks of intervention
  Percentage of dilatation of the brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Anil Nigam, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Cardiovascular Prevention and Rehabilitation Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Langeard A, Cloutier SO, Olmand M, Saillant K, Gagnon C, Gregoire CA, Fortier A, Lacroix M, Lalonge J, Gayda M, Besnier F, Gagnon D, Bherer L, Nigam A. High-intensity interval training vs. hydrochlorothiazide on blood pressure, cardiovascular health and cognition: Protocol of a non-inferiority trial. Contemp Clin Trials. 2021 Mar;102:106286. doi: 10.1016/j.cct.2021.106286. Epub 2021 Jan 20. PMID 33484896